CLINICAL TRIAL: NCT03741023
Title: Disorders of the Acute Phase Response Accelerated by Plasmin Activation Following Trauma and Invasive Surgery: A Prospective Study
Brief Title: Disorders of the Acute Phase Response Following Trauma and Invasive Surgery
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Jon Schoenecker, Associate Professor of Orthopaedic Surgery, Associate Professor of Pediatrics, Vanderbilt University Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 181982
Record Dates: First submitted 2018-10-31; First posted 2018-11-14 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Acute Phase Response
MeSH Terms: conditions — Acute-Phase Reaction | interventions — Blood Specimen Collection; Phlebotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Trauma Patients (Other): During Hospitalization:
  Patients routinely have blood drawn at time of admission and every 12 hours following admission up until 2 weeks post-admission or until discharge. Remnants of the blood draw will be stored in the Vanderbilt Lab core and retrieved for further analysis by key research personnel. Patients will have an additional 5.2ml of blood drawn (2 blue-top tubes) per time point during their normal course of care for this study, for a total of 72.8 mL of blood drawn per week. In addition to the routine blood draws, a finger stick may also be obtained the same day. Approximately 3 drops of blood (100μL maximum) will be removed by the finger stick.. Finger sticks will not be collected in the pediatric population.
  Follow-Up Visits Any complications resulting from traumatic injury will be documented at these routine care visits. These complications will be documented if they occur within 2 years of injury.
  Interventions: Procedure: Blood draw (venipuncture or fingerstick)
- Invasive Elective Surgery Patients (Other): During Hospitalization:
  Patients routinely have blood drawn pre-, intra- and post-operatively. Remnants of the blood draw will be stored in the Vanderbilt Lab core and retrieved for further analysis by key research personnel. Patients will have an additional 5.2ml of blood drawn (for patients 7 years of age or older) or 2mL of blood drawn (for patients under the age of 7 years old) immediately prior to surgery, every 30 minutes intraoperatively, every 6 hours for 3 days post-operatively, and every 12 hours from 3 days post-operative until discharge. Total blood volume drawn within one week will not exceed 150mL for patients ≥7 years of age and 55mL for patients <7 years of age (~3% total blood volume).
  Follow-Up Visits Any complications resulting from surgery will be documented at these routine care visits. These complications will be documented if they occur within 2 years of surgery.
  Interventions: Procedure: Blood draw (venipuncture or fingerstick)
- Healthy Volunteers (Other): Blood will be taken from healthy, non-pregnant adults who weigh at least 110 pounds by research staff trained in venipuncture at a one-time study visit.
  Interventions: Procedure: Blood draw (venipuncture or fingerstick)

INTERVENTIONS:
Procedure: Blood draw (venipuncture or fingerstick) — Blood will be drawn from participants by venipuncture and/or by fingerstick. Finger sticks will not be collected in the pediatric population.

SUMMARY:
The purpose of the proposed study is to test these hypotheses through the following aims:

1. To determine if early plasmin activation following severe injury correlates with SIRS, TIC and complications throughout convalescence in both trauma and surgical patients.
2. To determine if early plasmin activation following severe injury correlates with plasminogen consumption and poor plasmin activity later in convalescence.

DETAILED DESCRIPTION:
Significance: Severe injury is a leading cause of death and disability worldwide, affecting approximately 2.8 million individuals and accounting for over 200,000 deaths annually across the United States1,2,3. Large cohort studies have demonstrated that approximately 64% of trauma-related deaths are due to complications including thrombosis, bleeding, infection, and organ dysfunction, and each complication corresponds with an 8% increase in risk of mortality4. While advances in critical care medicine have significantly improved the initial survival from traumatic injuries, the proportion of morbidity and mortality from complications experienced during traumatic convalescence has correspondingly skyrocketed. Early in convalescence, these patients are at risk of developing life-threatening complications instigated by trauma induced coagulopathy (TIC) and systemic inflammatory response syndrome (SIRS). Specifically, approximately 40% of patients with severe injuries develop TIC and approximately 70% develop SIRS5,6. While these conditions individually increase the risk of secondary sequelae, in concurrence, they dramatically increase the risk of bleeding, thrombosis, infection, and multi-organ dysfunction syndrome (MODS)7,8,9. Later in convalescence, patients experiencing severe injury are at risk of suffering complications from pathologic tissue homeostasis and repair. For example, depending on the injury, 25-65% of severely injured patients' rehabilitation and quality of life are limited by poor bone health, including the development of osteoporosis, impaired bone healing, and/or the development of heterotopic ossification10,11,12. Together, early and late complications of convalescence reportedly account for over $671 billion in healthcare expenditure and disability losses yearly1. Thus, there is an unmet need for improved therapeutic and diagnostic measures for these patients to prevent or treat complications of early and late convalescence.

The Acute Phase Response (APR): Following injury, the APR resolves the four principle problems provoked by disruption of tissue: bleeding, pathogen invasion, tissue hypoxia, and tissue dysfunction. After an isolated injury, e.g., femur fracture, the APR follows a predictable and quantifiable time-course with minimal risk of complications (Figure 1A). The survival phase contains the injury and prevents infection through hemostasis (fibrin deposition) and acute inflammation. The later repair phase effectively removes damaged tissue, regenerates new tissue, and restores function. Severe trauma derails the survival-APR, provoking complications in both in early and late convalescence (Figure 1B). In order to prevent exsanguination, severe trauma must provoke an adequate survival-APR in proportion to the severity of the injury. However, unrestrained and prolonged activation of coagulation and survival-inflammation lead to the development of TIC and SIRS and significantly increasing the risk of bleeding, thrombosis, and MODS6,5,8. Additionally, if a patient persists within the survival-APR for an extended period of time, the prolonged activation of cellular inflammation promotes disorders of tissue homeostasis, e.g., osteoporosis, and delays the transition to the repair-APR, stalling or preventing healing tissue and crippling recovery in these patients13,14. Therefore, APR complications are mechanistically linked, that is, dysfunction of the survival-APR contributes to dysfunction of the repair-APR. Although there are many reports suggesting potential molecular determinants of a dysfunctional APR, the primary molecular targets driving this phenomenon are unknown.

Severe Trauma-Provoked Changes in Plasmin Activity: Plasmin is converted from its zymogen, plasminogen, by its activators: tissue plasminogen activator (tPA) and urokinase plasminogen activator (uPA). While plasmin is a multifunctional protease, its canonical role is the degradation of fibrin (fibrinolysis). While fibrinolysis occurs during the repair-APR following an isolated injury, a severe injury provokes early hyperactivation of plasmin (Figure 2)15,16. Fibrinolysis was first observed by anatomist Giovanni Morgagni and surgeon John Hunter in the late 1700s during autopsies of individuals that suffered traumatic injuries17,18. Both Morgagni and Hunter noted that blood from these individuals strangely did not clot. It was later determined that blood clots formed following traumatic injury or invasive surgery spontaneously dissolved, leading to the discovery of plasmin.

The immediate and most-recognized clinical consequence of this inappropriate hyperfibrinolysis is bleeding, as the degradation of fibrin opposes effective hemostasis19. The clinical significance of injury- induced hyperfibrinolysis was propelled by improvements in critical care medicine that permitted not only survival of previously fatal traumatic injuries, but also invasive, elective surgical procedures through the use of antifibrinolytic therapeutics. Specifically, recent clinical studies in >40,000 trauma patients have demonstrated that prevention of plasmin activation by antifibrinolytics (e.g., aminocaproic acid (Amicar), tranexamic acid (TXA)) significantly reduced blood loss and increased survival when administered early after injury20,21. Thus, it has been established that inappropriate, early plasmin activation (hyperfibrinolysis) is a significant cause of bleeding and mortality following severe injury19,16.

Pathologic Fibrinolysis - Hemorrhage is the Tip of the Iceberg: Both hyperfibrinolysis and hypofibrinolysis occur following trauma and have been associated with complications throughout convalescence22,23, indicating that plasmin's biologic role following injury is more complex than previously understood. Indeed, since the initial investigations of plasmin's role in bleeding, our knowledge of the biological role of plasmin has greatly expanded beyond its role in hemostasis. Currently, it is recognized that plasmin is activated during virtually all tissue repair, where it degrades intra- and extravascular fibrin24,25. In addition to fibrinolysis, plasmin also acts through non-canonical pathways to promote tissue repair including programming and migration of macrophages and progenitor cells, growth factor activation, and promotion of angiogenesis26,27,28,29. Additionally, plasmin stimulates an acute inflammatory response, promoting tissue regeneration30,31,32. Thus, plasmin is essential for tissue maintenance and repair. Specifically, our lab has extended this premise by determining that plasmin is essential for proper bone homeostasis, as well as bone and muscle repair33,34,35. Thus, following trauma, the biological role of plasmin is not limited to intravascular activity and bleeding. Instead, it plays well defined, albeit less understood, roles in pro- and anti-inflammatory responses, tissue homeostasis, and repair of virtually all tissues. While these studies would suggest that plasmin plays beneficial role in recovery following trauma, judicious prevention of early plasmin activation is clearly beneficial in preventing life threatening hemorrhage.

The purpose of the proposed study is to test these hypotheses through the following aims:

1. To determine if early plasmin activation following severe injury correlates with SIRS, TIC and complications throughout convalescence in both trauma and surgical patients.
2. To determine if early plasmin activation following severe injury correlates with plasminogen consumption and poor plasmin activity later in convalescence.

ELIGIBILITY:
Arm 1: Level I Trauma Patients Inclusion criteria

* Any patient admitted to or treated in the VUMC Adult Trauma Unit
* Patients ages 16 and older (all included in the adult trauma unit admissions)
* Patients will be divided into sub-groups for analyses based on type of trauma (TBI, blunt force trauma, polytrauma, etc) and severity (Level 1 vs non-level 1 trauma)

Exclusion criteria

• None

Arm 2: Invasive Elective Surgical Patients Inclusion criteria

* Any patient admitted for an invasive elective surgery associated with high blood loss or a high risk of vascular complications at VUMC/VCH. Enrollment will be at the discretion of the attending physician
* This may include, but is not limited to, orthopedic and vascular surgery patients
* Patients ages 2 months and older Exclusion criteria
* None

Arm 3: Healthy Volunteers Inclusion criteria

* Volunteers should be male or female
* Age 18-70 years of age
* Weight greater than 110lbs

Exclusion criteria

* Chronic medical conditions such as: diabetes, hypertension, high cholesterol, rheumatologic disorders, infections, etc.
* No history of recent traumatic injury (within the past year)
* Pregnant females or people on hormone replacement therapy
* People on any anticoagulant medication or NSAIDS

Min Age: 2 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2019-12-12 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Interleukin-6 (IL-6) | During hospitalization (approximately 7-21 days)
  A change in Interleukin-6 (IL-6) lab value following traumatic injuries or traumatic elective surgeries will be used to determine change in systematic inflammation.
Thrombin-Antithrombin (TAT) Complex | During hospitalization (approximately 7-21 days)
  A change in the Thrombin-antithrombin (TAT) complex following traumatic injuries or traumatic elective surgeries will be used to determine change in coagulation.
D-Dimer | During hospitalization (approximately 7-21 days)
  A change in d-dimer lab value following traumatic injuries or traumatic elective surgeries will be used to determine change in fibrinolysis.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Schoenecker, MD, PhD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt Univeristy Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gibson BHY, Duvernay MT, McKeithan LJ, Benvenuti TA, Warhoover TA, Martus JE, Mencio GA, Emerson BR, Moore-Lotridge SN, Borst AJ, Schoenecker JG. Variable Response to Antifibrinolytics Correlates with Blood-loss and Transfusion in Posterior Spinal Fusion. Spine Deform. 2022 Jul;10(4):841-851. doi: 10.1007/s43390-022-00489-6. Epub 2022 Mar 5. PMID 35247191

DOCUMENTS (1):
  • Informed Consent Form (2021-04-12): https://cdn.clinicaltrials.gov/large-docs/23/NCT03741023/ICF_003.pdf